CLINICAL TRIAL: NCT04839146
Title: First-in-human Trial of the Coronavirus Virus-like Particle Subunit Vaccine ABNCoV2 in SARS-CoV-2-naïve Adult Volunteers in Good Health
Brief Title: Safety and Tolerability of COVID-19 Vaccine (ABNCoV2)
Acronym: COUGH-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL76192.000.20
Record Dates: First submitted 2021-03-11; First posted 2021-04-09 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Severe Acute Respiratory Syndrome; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — ABNCoV2 vaccine

STUDY DESIGN:
Intervention Model Description: ABNCoV2 is a virus-like particle vaccine. It will be administered as two intramuscular injections in groups of up to 9 volunteers. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination. The pre-defined escalation schedule will start with 6 μg ABNCoV2, followed by 12, 25 and 50 μg with a maximum dose of 70 μg. MF59-adjuvanted and non-adjuvanted formulations will be tested in parallel to detect superiority or futility of the MF59-adjuvanted against the non-adjuvanted formulation at the 6, 12 and 25 μg dosage. Approval for further dose escalation and choice of adjuvant use will be provided by a safety monitoring committee (SMC), supported by pre-defined analyses of safety, tolerability and immunogenicity data at day 14 post-first-vaccination. Recruitment for the two best (safe, tolerable and most immunogenic) regimens will continue until 12 volunteers per regimen have been immunized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1: 6 microgram ABNCoV2 with/without MF59 adjuvant (Experimental): In Group 1 (n=6), subjects will receive 6 μg ABNCoV2 intramuscularly, half of whom (n=3) will receive the non-adjuvanted vaccine formulation and the other half (n=3) will receive the MF59-adjuvanted vaccine formulation. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine
- Group 2: 12 microgram ABNCoV2 with/without MF59 adjuvant (Experimental): In Group 2 (n=6), subjects will receive 12 μg ABNCoV2 intramuscularly, half of whom (n=3) will receive the non-adjuvanted vaccine formulation and the other half (n=3) will receive the MF59-adjuvanted vaccine formulation. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine
- Group 3: 25 microgram ABNCoV2 with/without MF59 adjuvant (Experimental): In Group 3 (n=6), subjects will receive 25 μg ABNCoV2 intramuscularly, half of whom (n=3) will receive the non-adjuvanted vaccine formulation and the other half (n=3) will receive the MF59-adjuvanted vaccine formulation. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine
- Group 4: 50 microgram ABNCoV2 with/without MF59 adjuvant (Experimental): In Group 4 (n=6), subjects will receive 50 μg non-adjuvanted or MF59-adjuvanted ABNCoV2 intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine
- Group 5: 70 microgram ABNCoV2 with/without MF59 adjuvant (Experimental): In Group 5 (n=6), subjects will receive 70 μg non-adjuvanted or MF59-adjuvanted ABNCoV2 intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine
- Group 6: t.b.d. microgram ABNCoV2 with/without MF59 adjuvant (Experimental): The subjects in Group 6 (n=6) will receive the next lower dosage of the highest non-adjuvanted or MF59-adjuvanted ABNCoV2 dose achieved intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine
- Group 7: t.b.d. microgram ABNCoV2 with/without MF59 adjuvant (Experimental): The subjects in Group 7 (n=6) will receive the highest non-adjuvanted or MF59-adjuvanted ABNCoV2 dose achieved intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  Interventions: Biological: ABNCoV2 Vaccine

INTERVENTIONS:
Biological: ABNCoV2 Vaccine — SARS-CoV-2 vaccine
  Other Names: cVLP-RBD; RBDn-CLP; ABNCoV2

SUMMARY:
This phase 1 trial aims to assess the safety and tolerability of two doses of ABNCoV2, formulated with and without the adjuvant MF59, in healthy adult volunteers and to identify the dosage and formulation that optimizes the immunogenicity-tolerability ratio 14 days following first vaccination with ABNCoV2.

DETAILED DESCRIPTION:
This first-in-human phase 1 trial of ABNCoV2 is a single center, sequential dose-escalation, open labelled trial to establish the safety and tolerability of two doses of ABNCoV2, formulated with and without MF59 in healthy, adult, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-naïve volunteers. The immunological objective of this trial is to identify a dosage that optimizes the immunogenicity-tolerability ratio 14 days following first vaccination with ABNCoV2. The trial will be carried out by the Radboud University Medical Center (Radboudumc).

The trial involves first-in-human administration, dose escalation of ABNCoV2 and adjuvant selection. Volunteers will be screened for eligibility and receive two vaccinations by intramuscular injection. While we cannot predict with certainty the safety in human subjects, we have adopted a safety-orientated staggered trial design with ascending doses of ABNCoV2. Seven groups of volunteers (n=6) will receive a given dose of ABNCoV2, either with or without MF59, followed by a booster with the same dose and formulation four weeks after the first vaccination. All vaccinations will be given as intramuscular injection. The pre-defined escalation schedule will start with 6 μg ABNCoV2, with a maximum dose of 70 μg. Dose-escalation will proceed only in absence of protocol-defined safety signals. MF59-adjuvanted and non-adjuvanted formulations will be tested in parallel at the first three escalation steps (Group 1-3) to detect superiority or futility of the MF59-adjuvanted against the non-adjuvanted formulation. Up to forty-two (n=42) subjects will be enrolled, as well as one reserve subject per group.

Safety follow-up will be done at following timepoints: baseline, day 1, day 2, day 7, day 14, day 25, day 29, day 30, day 35, day 42, day 70, day 119 and day 196 after first ABNCoV2 administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign written informed consent to participate in the trial.
2. Subject is able to understand planned study procedures and demonstrate comprehension of the protocol procedures and knowledge of the study by passing a quiz (assessment of understanding). Subjects must score at least 80% correct on a multiple-choice quiz. If they do not score 80% on the initial quiz, the protocol information will be reviewed with them, and they will have the opportunity to retest.
3. In the opinion of the investigator, the subject can and will comply with the requirements of the protocol.
4. Subjects are available to attend all study visits and are reachable by phone throughout the entire study period from day -1 until 24 weeks following last vaccination (end of study).
5. Subject is a male or non-pregnant and non-lactating female age ≥ 18 and ≤ 55 years and in good health at time of ABNCoV2 administration.
6. Subject agrees to their general practitioner (GP) being informed about participation in the study and agrees to sign a form to request the release by their GP, and medical specialist when necessary, of any relevant medical information concerning possible contra-indications for participation in the study to the investigator(s).
7. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period according to current Sanquin guidelines.
8. Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause. All other female subjects must agree to use continuous adequate contraception2 for the duration of the study. Female subjects must have a negative pregnancy test at the inclusion visit.

Exclusion Criteria:

Any clinically significant abnormal finding on clinical examination or laboratory screening tests according to the US Food and Drug Administration (FDA) Toxicity Grading Scale for Healthy Adult and Adolescent Subjects Enrolled in Preventative Vaccine Clinical Trials [30].

2. History of COVID-19 infection. 3. Chronic use of immunosuppressive drugs or other immune modifying drugs within six months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

4. Positive urine toxicology test for cannabis, cocaine or amphetamines at inclusion.

5. Screening tests positive for SARS-CoV-2, SARS-CoV-2 antibodies, Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV).

6. Receipt of any investigational or non-registered product (drug or vaccine) other than the study product in the 30 days preceding enrolment or during the study period.

7. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.

8. Immunization with any vaccines within the past four weeks or planned receipt of a vaccine during the study period with the exception of a licensed SARS-CoV-2 vaccine, given within the framework of the national SARS-CoV-2 vaccination campaign. The time between last vaccination with ABNCoV2 and a SARS-CoV-2 vaccine provided by the campaign shall be at least 4 weeks.

9. Known hypersensitivity to any of the vaccine components (adjuvant or protein).

10. Administration of immunoglobulins and/or any blood products within the three months prior to the first dose of ABNCoV2 or planned administration during the study period.

11. Previous participation in a COVID-19 vaccine study. 12. Body Mass Index (BMI) >35 kg/m2. 13. Pregnancy, lactation or intention to become pregnant during the study period.

14. History of drug or alcohol abuse interfering with normal functioning in the five years preceding enrolment.

15. Being an employee or student of the department of Medical Microbiology of the Radboudumc, or a person otherwise related to the investigator other than a professional relationship for clinical trial purpose only.

16. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Mordmüller, Prof, Principal Investigator — Stichting Radboud university medical center
Locations (1):
- Radboud univserity medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Smit MJ, Sander AF, Ariaans MBPA, Fougeroux C, Heinzel C, Fendel R, Esen M, Kremsner PG, Ter Heine R, Wertheim HF, Idorn M, Paludan SR, Underwood AP, Binderup A, Ramirez S, Bukh J, Soegaard M, Erdogan SM, Gustavsson T, Clemmensen S, Theander TG, Salanti A, Hamborg M, de Jongh WA, McCall MBB, Nielsen MA, Mordmuller BG; COUGH-1 trial study group. First-in-human use of a modular capsid virus-like vaccine platform: an open-label, non-randomised, phase 1 clinical trial of the SARS-CoV-2 vaccine ABNCoV2. Lancet Microbe. 2023 Mar;4(3):e140-e148. doi: 10.1016/S2666-5247(22)00337-8. Epub 2023 Jan 18. PMID 36681093

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant; Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant: In Group 1 (n=6), subjects will receive 6 μg ABNCoV2 intramuscularly, half of whom (n=3; Group 1A) will receive the non-adjuvanted vaccine formulation and the other half (n=3; Group 1B) will receive the MF59-adjuvanted vaccine formulation. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
- Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant; Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant: In Group 2 (n=6), subjects will receive 12 μg ABNCoV2 intramuscularly, half of whom (n=3; Group 2A) will receive the non-adjuvanted vaccine formulation and the other half (n=3; Group 2B) will receive the MF59-adjuvanted vaccine formulation. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
- Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant; Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant: In Group 3 (n=6), subjects will receive 25 μg ABNCoV2 intramuscularly, half of whom (n=3; Group 3A) will receive the non-adjuvanted vaccine formulation and the other half (n=3; Group 3B) will receive the MF59-adjuvanted vaccine formulation. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
- Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant: In Group 4 (n=6), subjects will receive 50 μg non-adjuvanted ABNCoV2 intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
- Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant: In Group 5 (n=6), subjects will receive 70 μg non-adjuvanted ABNCoV2 intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
- Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant: The subjects in Group 6 (n=9) will receive 25 μg non-adjuvanted ABNCoV2 intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
- Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant: The subjects in Group 7 (n=6) will receive 50 μg non-adjuvanted ABNCoV2 intramuscularly. All subjects will receive a second vaccination with the same dose and formulation 4 weeks following the first vaccination.
  ABNCoV2 Vaccine: SARS-CoV-2 vaccine
Period: Overall Study
Arm/Group | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant
Started | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 9 | 6
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 9 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 9 | 6 | 45
Age, Continuous [Median (Full Range); unit: years] | 31 [21 to 35] | 27 [22 to 52] | 25 [23 to 34] | 37 [22 to 37] | 27 [22 to 28] | 48 [33 to 54] | 25.5 [20 to 44] | 20.5 [20 to 46] | 24 [21 to 45] | 24 [18 to 29] | 26 [18 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 2 | 4 | 3 | 4 | 3 | 26
  Male | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 3 | 5 | 3 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Bodyweight (kg) [Median (Full Range); unit: kg] | 79 [61 to 96] | 66 [59 to 69.6] | 78 [76 to 89.4] | 88 [62 to 94] | 70.1 [61.2 to 79] | 81 [72.8 to 91] | 75 [60 to 97] | 77.5 [66 to 90] | 76.6 [61 to 91] | 69.5 [60 to 88] | 76 [59 to 97]
BMI (kg/m2) [Median (Full Range); unit: kg/m2] | 23 [22.1 to 31.0] | 22.4 [18.4 to 24.4] | 26.0 [24.9 to 32.1] | 24.9 [22.8 to 28.4] | 23.6 [20.5 to 25.4] | 26.4 [24.9 to 26.9] | 25.0 [17.5 to 27.3] | 23.7 [20.5 to 26.6] | 23.3 [20.4 to 29.9] | 24.5 [20.5 to 27.1] | 24.2 [17.5 to 32.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of at Least Possibly Related Grade 3 Adverse Events (AE) and Serious Adverse Events (SAE)
Description: Primary safety endpoint: Number of at least possibly related Grade 3 adverse events (AE) and serious adverse events (SAE)
Time Frame: up to 28 weeks
Measure: Number; unit: adverse events
Arm/Group | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 9 | 6
adverse events | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Concentration of ABNCoV2-specific Antibodies 14 Days Following First Vaccination
Description: Primary immunogenicity endpoint: Concentration of ABNCoV2-specific antibodies 14 days following first vaccination
Time Frame: 14 days following first vaccination.
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 9 | 6
ug/mL | 2.2 [0.4 to 5.8] | 4.9 [3.6 to 30.1] | 7.1 [2.3 to 7.1] | 9.4 [8.7 to 95.5] | 2.3 [1.6 to 34.4] | 0.4 [0.4 to 5.7] | 4.2 [2.4 to 22.0] | 4.9 [0.1 to 16.8] | 5.0 [1.7 to 20.4] | 7.3 [5.5 to 35.1]

3. Secondary Outcome: Number and Severity of at Least Possibly Related Solicited AEs
Description: Secondary study endpoint: Number and severity of at least possibly related solicited AEs
Time Frame: within one week following administration of ABNCoV2.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Concentration of ABNCoV2-specific Antibodies at Baseline and During Immunization and Follow up.
Description: ABNCoV2-specific antibody concentrations will be measured by ELISA during immunisation and follow-up.
Time Frame: up to 28 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Inhibitory Titre in Invasion Inhibition Assay at Baseline and During Immunization and Follow up.
Description: Inhibitory titre in invasion inhibition assay at baseline and during immunization and follow up. Inhibitory titres will be measured in an in vitro SARS-CoV-2 invasion inhibition assay.
Time Frame: up to 28 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cellular Immune Responses (T and B Cell) at Baseline and During Immunization and Follow up.
Description: Cellular responses will be analysed by cytometry and enzyme-linked absorbent spot (ELISpot) assay.
Time Frame: up to 28 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Correlation of Response Vaccine to Habitual Sleep Using the Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI will be used to investigate if sleep quality is associated with immune responses to the vaccine.
Time Frame: one month prior first ABNCoV2 immunization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/9 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 6/6 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant (N=3) | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant (N=3) | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant (N=3) | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant (N=3) | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant (N=3) | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant (N=3) | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant (N=6) | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant (N=6) | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant (N=9) | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant (N=6)
Superficial basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Traumatic ligament rupture requiring hospitalisation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A: 6 Microgram ABNCoV2 Without MF59 Adjuvant (N=3) | Group 1B: 6 Microgram ABNCoV2 With MF59 Adjuvant (N=3) | Group 2A: 12 Microgram ABNCoV2 Without MF59 Adjuvant (N=3) | Group 2B: 12 Microgram ABNCoV2 With MF59 Adjuvant (N=3) | Group 3A: 25 Microgram ABNCoV2 Without MF59 Adjuvant (N=3) | Group 3B: 25 Microgram ABNCoV2 With MF59 Adjuvant (N=3) | Group 4: 50 Microgram ABNCoV2 Without MF59 Adjuvant (N=6) | Group 5: 70 Microgram ABNCoV2 Without MF59 Adjuvant (N=6) | Group 6: 25 Microgram ABNCoV2 Without MF59 Adjuvant (N=9) | Group 7: 50 Microgram ABNCoV2 Without MF59 Adjuvant (N=6)
Tenderness (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 3 (3) | 2 (3) | 1 (2) | 3 (6) | 5 (8) | 3 (5) | 8 (11) | 3 (4) — Tenderness at injection site (solicited local adverse event)
Pain (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 3 (7) | 3 (6) | 3 (7) | 3 (9) | 5 (21) | 6 (15) | 9 (21) | 6 (14) — Pain at injection site (solicited local adverse event)
Induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 4 (4) | 3 (3) — Induration at injection site (solicited local adverse event)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 2 (3) | 3 (3) — Erythema at injection site (solicited local adverse event)
Chills (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 1 (1) | 1 (1) | 2 (3) — Chills (solicited systemic adverse event)
Drowsiness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4) — Drowsiness (solicited systemic adverse event)
Fatigue (General disorders) | 1 (1) | 2 (4) | 2 (3) | 3 (4) | 0 (0) | 2 (7) | 4 (6) | 3 (6) | 6 (9) | 4 (5) — Fatigue (solicited systemic adverse event)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) — Fever (solicited systemic adverse event)
Headache (General disorders) | 1 (1) | 3 (6) | 2 (2) | 2 (3) | 3 (3) | 2 (5) | 4 (7) | 2 (7) | 6 (9) | 3 (4) — Headache (solicited systemic adverse event)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT04839146/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT04839146/SAP_001.pdf